CLINICAL TRIAL: NCT05804214
Title: Observational Study of Infants Fed With Dairy and Plant Based Infant Formula
Acronym: Complement
Status: Terminated | Type: Observational
Why Stopped: Study early terminated
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SBB22R&41357
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Infant Growth; Parent and Infant User Experience
Keywords: Complement; infant formula; dairy and plant based

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants who started feeding with the product at ≤ 4 months of age: Infants who started feeding with the product at ≤ 4 months of age, either supplemental to breastfeeding or as sole source of feeding
  Interventions: Other: Dairy and plant based infant formula feeding

INTERVENTIONS:
Other: Dairy and plant based infant formula feeding — Parents have already decided to feed their infant with the product (a dairy and plant based infant formula) daily, starting within the first 4 months of life, continuing for at least 2 months

SUMMARY:
A study to assess and evaluate adequate growth in infants receiving a dairy and plant based infant formula in a real-world setting, and parents' and infants' experiences with this infant formula.

DETAILED DESCRIPTION:
The study collects growth data from 58 participating infants whose parents autonomously decided to use the dairy and plant based infant formula for their infant daily within the first three months of their infant's life, either supplemental to breastfeeding or as sole source of feeding. Parents are asked to complete 2-3 online questionnaires in which data is collected on infant growth (as assessed during regular visits to the Municipal Child Healthcare Clinic), feeding characteristics, parent and infant experience with the product, and whether their infant has been to a doctor or is taking medication.

ELIGIBILITY:
Inclusion Criteria:

1. Parents autonomously decided to feed their infant with at least one bottle per day of dairy and plant based infant formula in combination with breastfeeding or as sole source of feeding.
2. Parents' intention to feed their infant with dairy and plant based infant formula for at least 2 months as of start with product
3. Infant started feeding with dairy and plant based infant formula ≤ 4 months of age
4. Infant is being fed daily with dairy and plant based infant formula at time of enrolment

Exclusion Criteria:

1. Infant started feeding with dairy and plant based infant formula >3 months ago at time of enrolment
2. Participation of the infant in any other studies involving infant formula feeding (products) concomitantly

Max Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants that are fed with dairy and plant based infant formula ≤ 4 months of age. Infants should be enrolled within three months after start with dairy and plant based infant formula.
  Before screening, parents should already autonomously have decided to use dairy and plant based infant formula for their infant according to the label of the product.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Development of weight, length, and head circumference | 5 Months +2 weeks
  Agreed clinical experts' judgement about development of weight, length and head circumference (adequate/inadequate) as measured at the Municipal Child Healthcare Clinic visits and transcribed by the parents in a digital tool

SECONDARY OUTCOMES:
Development of length, BMI, and head circumference | 5 Months + 2 weeks
  Agreed clinical experts' judgement about adequate development of length, BMI (derived from weight and length outcomes), and head circumference (adequate/inadequate)
Weight-for-age, length-for-age, BMI-for-age, and head circumference-for-age | 5 Months + 2 weeks
  Weight-for-age, length-for-age, BMI-for-age, and head circumference-for-age since start of the dairy and plant based infant formula (according to the country specific z-score by age and sex)
Experience of parent and infant | after using product for 2 and 5 Months
  Parent's and infant's experiences with the dairy and plant based infant formula after using the product for 2 and 5 months and assessed via a digital questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Ncru, Danone Nutricia Research, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided